CLINICAL TRIAL: NCT04111926
Title: Impact of Intraoperative Dexmedetomidine on Long-term Outcomes in Elderly Patients After Major Non-cardiac Surgery: 3-year Follow-up of a Randomised Controlled Trial
Brief Title: Intraoperative Dexmedetomidine and Long-term Outcomes in Elderly After Major Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-0927
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Overall Survival
Keywords: Elderly patients; Major non-cardiac surgery; Dexmedetomidine; long-term survival
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A loading dose of dexmedetomidine (0.6 μg/kg) was administered during a 10-minute period before anaesthesia induction, followed by a continuous infusion at a rate of 0.5 μg/kg/hr till 1 hour before the end of surgery.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): Volume-matched normal saline was administered in the same rate for the same duration as in the intervention group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — A loading dose of dexmedetomidine (0.6 μg/kg) was administered during a 10-minute period before anaesthesia induction, followed by a continuous infusion at a rate of 0.5 μg/kg/hr till 1 hour before the end of surgery.
  Other Names: Dexmedetomidine Hydrochloride
  Arms: Intervention group
Drug: Placebo — Volume-matched normal saline was administered in the same rate for the same duration as in the intervention group.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
This is a 3-year follow-up of patients enrolled in a previous randomized controlled trial which showed that intraoperative dexmedetomidine reduced delirium in elderly patients after major non-cardiac surgery. The purpose of this study is to clarify the effects of intraoperative dexmedetomidine on long-term outcomes of these patients.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective α-2-receptor agonist with sedative, analgesic and anxiolytic effects. When used as an supplement during general anaesthesia, it reduces the consumption of the anaesthetics and relieves surgery-related stress response and inflammation. In a recent randomized ontrolled trial of the applicants, 620 elderly patients who underwent major non-cardiac surgery were randomized to receive dexmedetomidine or normal saline during general anesthesia. The results showed that use of dexmedetomidine reduced delirium (5.5% [17/309] with dexmedetomidine vs. 10.2% [32/310] with placebo, P=0.026) and 30-day non-delirium complications (9.4% [60/309] with dexmedetomidine vs. 26.1% [81/310] with placebo, P=0.047) after surgery.

The effects of intraoperative dexmedetomidine on long-term outcomes after surgery remains unclear. In another study of the applicants, use of low-dose dexemeditomidine in ICU patients after surgery increased survival up to 2 years and improve quality of life in 3-year survivors. On the contrary, it was reported in a retrospective study that intraoperative use of dexmedetomidine was associated with shortened overall survival in patients after lung cancer surgery. Therefore, it is urgent to clarify the impact of intraoperative dexemeditomidine on long-term outcomes of patients undergoing major surgery, especially those undergoing cancer surgery.

This study is a 3-year follow-up of patients who were enrolled in a randomzied controlled trial of the applicants in order to clarify the effects of intraoperative dexmedetomidine on long-term outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age ≥60 years);
* Scheduled to undergo elective major non-cardiac surgery with expected duration ≥2 hours under general anaesthesia.

Exclusion Criteria:

* Do not provide written informed consent;
* Previous history of schizophrenia, epilepsy or Parkinson's disease;
* Visual, hearing, language or other barriers which impede communication and preoperative delirium assessment;
* History of traumatic brain injury;
* Severe bradycardia (heart rate <40 beats per minutes), sick sinus syndrome, or atrioventricular block of degree 2 or above without pacemaker;
* Severe hepatic dysfunction (Child-Pugh grade C);
* Renal failure (requirement of renal replacement therapy);
* Neurosurgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Overall survival within 3 years after surgery | Up to 3 years after surgery.
  Overall survival within 3 years after surgery

SECONDARY OUTCOMES:
Recurrence-free survival within 3 years after surgery. | Up to 3 years after surgery.
  Recurrence-free survival within 3 years after surgery.
Cancer-specific survival within 3 years after surgery. | Up to 3 years after surgery.
  Cancer-specific survival within 3 years after surgery.
Rate of new-onset disease or hospital readmission within 3 years after surgery. | Up to 3 years after surgery.
  Rate of new-onset disease or hospital readmission within 3 years after surgery.
Quality of life in 3-year survivors. | At 3 years after surgery.
  Quality of life is assessed with the World Health Organization Quality of Life-Brief Version. It assesses the quality of life at 4 domains, i.e., physical, psychological, social relationships, and environment. The score of each domain ranges from 0 to 100, with higher score indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Meguid ME. Dexmedetomidine as anesthetic adjunct for fast tracking and pain control in off-pump coronary artery bypass. Saudi J Anaesth. 2013 Jan;7(1):6-8. doi: 10.4103/1658-354X.109557. PMID 23717223
- [Background] Jalonen J, Hynynen M, Kuitunen A, Heikkila H, Perttila J, Salmenpera M, Valtonen M, Aantaa R, Kallio A. Dexmedetomidine as an anesthetic adjunct in coronary artery bypass grafting. Anesthesiology. 1997 Feb;86(2):331-45. doi: 10.1097/00000542-199702000-00009. PMID 9054252
- [Background] Li Y, Wang B, Zhang LL, He SF, Hu XW, Wong GT, Zhang Y. Dexmedetomidine Combined with General Anesthesia Provides Similar Intraoperative Stress Response Reduction When Compared with a Combined General and Epidural Anesthetic Technique. Anesth Analg. 2016 Apr;122(4):1202-10. doi: 10.1213/ANE.0000000000001165. PMID 26991622
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Wang BJ, Li CJ, Hu J, Li HJ, Guo C, Wang ZH, Zhang QC, Mu DL, Wang DX. Impact of dexmedetomidine infusion during general anaesthesia on incidence of postoperative delirium in elderly patients after major non-cardiac surgery: study protocol of a randomised, double-blinded and placebo-controlled trial. BMJ Open. 2018 Apr 21;8(4):e019549. doi: 10.1136/bmjopen-2017-019549. PMID 29680809
- [Background] Cata JP, Singh V, Lee BM, Villarreal J, Mehran JR, Yu J, Gottumukkala V, Lavon H, Ben-Eliyahu S. Intraoperative use of dexmedetomidine is associated with decreased overall survival after lung cancer surgery. J Anaesthesiol Clin Pharmacol. 2017 Jul-Sep;33(3):317-323. doi: 10.4103/joacp.JOACP_299_16. PMID 29109628
- [Background] Gerresheim G, Schwemmer U. [Dexmedetomidine]. Anaesthesist. 2013 Aug;62(8):661-74. doi: 10.1007/s00101-013-2206-6. German. PMID 23917892
- [Derived] Xing MW, Li CJ, Guo C, Wang BJ, Mu DL, Wang DX. Effect of intraoperative dexmedetomidine on long-term survival in older patients after major noncardiac surgery: 3-year follow-up of a randomized trial. J Clin Anesth. 2023 Jun;86:111068. doi: 10.1016/j.jclinane.2023.111068. Epub 2023 Feb 1. PMID 36736209